CLINICAL TRIAL: NCT01473823
Title: Treatment of IgE Associated Eczema With Omega-3 Long Chain Polyunsaturated Fatty Acids in Infancy and the Development of Bronchial Asthma in Childhood
Acronym: Omega-Treat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Karel Duchén, MD, Principal Investigator, Ostergotland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OT-013
Record Dates: First submitted 2011-11-09; First posted 2011-11-17 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Food Allergy; Eczema; Sensitisation
Keywords: food allergy; eczema; sensitisation; omega-3 long chain polyunsaturated fatty acids; prevention; asthma
MeSH Terms: conditions — Food Hypersensitivity; Eczema; Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo oil (Placebo Comparator): Canola oil with high oleic acid content flavored with lemon supplied as 5 ml daily.
  Interventions: Dietary Supplement: Omega-3 LCPUFA
- Omega-3 LCPUFA (Active Comparator): The omega-3 LCPUFA supplementation comprises of 5 ml daily of "Möller's Tran" flavored with lemon. This dose provides the child with 1200 mg of omega-3 fatty acid of which 600 mg is DHA and 400 mg is EPA.
  Interventions: Dietary Supplement: Omega-3 LCPUFA

INTERVENTIONS:
Dietary Supplement: Omega-3 LCPUFA — Dosage is 5 ml daily until age 3 years.

SUMMARY:
Although some causal factors in allergy development such as allergen exposure and environmental pollution have decreased during recent years, the incidence of the allergic diseases has increased in the Western world. Since the genetic predisposition to develop allergies cannot change in such a short time it is conceivable that, instead of the emerging of some new and unknown risk factors, some protective factors seem to have disappeared in the Western world.

Allergic disease is a tendency to develop allergies to allergens in the surrounding environment. The most common symptoms are eczema and food allergy in the early life, bronchial asthma (AB) later in childhood and allergic rhino conjunctivitis (ARC) during school age and adolescence, the so-called allergic march. Some person may develop only one, but others some or all of the symptoms. Inheritance, environment and allergen exposure are important factors affecting this march but there are important factors that predict later development of diseases. Sensitization to egg (positive skin prick test or specific IgE to egg in the serum) combined with skin problems in infancy predispose strongly to the development of allergic asthma in later life.

The purpose of this work is to supply children with early development of IgE associated eczema and food allergy with omega-3 LCPUFA before the age of 12 months and assess the effect of the supplementation on the future development of skin symptoms, food allergy, sensitisation against inhalant allergens and asthma in these children. We will also assess immunological markers of Th2-skewed immunity in relation to clinical effect of the supplementation.

Families with children younger than 12 months referred to the paediatric department at Linköping University Hospital, Motala, Norrköping and Jönköping Hospitals in the South East of Sweden, with the diagnosis IgE associated eczema and sensitised against food allergens (egg, milk, wheat and/or soya) will be invited to participate in this study. Clinical examination by a paediatrician and assessment of disease severity with SCORAD will be performed by a research nurse at inclusion. The children will be assessed every six months by a nurse until 2.5 years of age and by a paediatrician at 3 years of age. Later clinical assessment will be performed yearly until age 7.

ELIGIBILITY:
Inclusion Criteria:

* Eczema and sensitisation to food allergens

Exclusion Criteria:

* Fish allergy within family

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of bronchial asthma | 7 years

SECONDARY OUTCOMES:
Severity of allergic symptoms and sensitisations to inhalants | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Karel Duchén, MD, PhD, Principal Investigator — Ostergotland CC
Locations (1):
- Allergicentrum, Linköping, Sweden